CLINICAL TRIAL: NCT03732417
Title: Effectiveness of a Telematic Model Integrated in the Transversal Care of the Secondary Prevention of Patients With Stroke
Brief Title: Telematic Model Integrated in the Transversal Care of the Secondary Prevention of Patients With Stroke
Status: Withdrawn | Type: Observational
Why Stopped: The start of the study was temporarily interrupted due to the COVID-19 pandemic. Subsequently, it was not feasible to initiate the study due to changes in the healthcare system for patient follow-up. For this reason, the study was withdrawn.
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Sponsor
Other Study IDs: CEIC P18/071
Record Dates: First submitted 2018-10-05; First posted 2018-11-06 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Risk Factor, Cardiovascular
Keywords: Nurse's Role; quality of life; adherence; risk factors; stroke; secondary prevention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients: Control group included people with ischemic or haemorragic stroke in Terres de l'Ebre, Spain.
- Telematic model treatment of patients with Stroke: The intervention group included control and education for the patient's health to promote self-care and empowerment, and enhance pharmacological compliance. The telematic model has been developed through clinical practice guides of primary care and the most recent publications on the subject referenced.
  Interventions: Other: Secondary prevention of cardiovascular risk factors

INTERVENTIONS:
Other: Secondary prevention of cardiovascular risk factors — Intervention group (n=35) Control group (n=35)
  Groups: Telematic model treatment of patients with Stroke

SUMMARY:
In Spain, stroke is the leading cause of death in women and disability in adults, which is why it is currently one of the most important public health problems. It is known that the main cause of stroke is the lack of control of cardiovascular risk factors (CRF). Strategies have been diversified for patients with severe neurological involvement, while those without or with mild involvement, susceptible to repeat a stroke, have a very heterogeneous approach.

Objective: Design, implement and evaluate the effectiveness of the transversal telematic model of secondary prevention in patients who have suffered a stroke.

Methodology: Randomized clinical trial with a control group, open and multicentre. A total of 70 patients (35 per group) will be included who meet all the inclusion criteria and none of exclusion, attended by an acute stroke in the Hospital Verge de la Cinta de Tortosa. Variables: sociodemographic and clinical, FRC, stage of change, therapeutic compliance and CV. Outcome variables: impact of the stroke using the scale (SIS-16); control of CRF, new vascular events and mortality at 3, 6, 12, 18 and 24 months, integrable in the practice and computerized clinical history (HCI). Interventions: control and education for the patient's health to promote self-care and empowerment, and enhance pharmacological compliance. The telematic model has been developed through clinical practice guides of primary care and the most recent publications on the subject referenced. Export of data directly from the HCI.

Analysis of results with the SPSS 23.0 program, using regression and survival models.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years old, diagnosed of established ischemic stroke and / or TIA and attended by the HTVC neurology service, on discharge from home and with habitual residence in the Ebro Lands to be able to follow up .
* Informed consent of the signed study.

Exclusion Criteria:

* Patients suffering from other neurological injuries that interfere with the follow-up (established strokes, with or without MCA deviation, glioblastomas, etc.), life expectancy <6 months, modified Rankin scale score (MRS) ≥3 and present language barrier and / or aphasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Calculated for two independent samples, variable SIS stroke impact scale result (DS 1.6). Accepting an alpha risk of 0.05 and a beta risk of less than 0.2 in a bilateral contrast, 35 subjects are needed in the first group and 35 in the second to detect a difference equal to or greater than 0.18 units. It is assumed that the common standard deviation is 0.25. A tracking loss rate has been estimated of 10%.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Stroke Impact Scale | At the beginning of the enrollment, 3, 6 ,12, 18 and 24 months later.
  Change from Baseline The Stroke Impact Scale for disability at 3, 6, 12, 18 and 24 months. Score range [16-80].

CONTACTS AND LOCATIONS:
Locations (1):
- Silvia Reverté, Tortosa, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No